CLINICAL TRIAL: NCT01782573
Title: The Efficacy of Pre - Disinfection Skin Scrub With 4% Chlorhexidine Gluconate in Preventing Surgical Site Infections for Patients With Hepatectomy
Brief Title: The Efficacy of Chlorhexidine Gluconate Pre - Disinfection Scrubbing in Preventing Surgical Site Infections for Hepatectomy Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, Chen Yao - Li, MD, Changhua Christian Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CCH - 110801
Record Dates: First submitted 2013-01-29; First posted 2013-02-04 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: Liver Tumors
Keywords: pre - disinfection scrubbing solution; surgical site culture; surgical site infection; liver tumors; hepatectomy; chlorhexidine gluconate
MeSH Terms: conditions — Carcinoma, Hepatocellular; Surgical Wound Infection | interventions — chlorhexidine gluconate; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chlorhexidine gluconate ( CHG ) (Active Comparator): (i)a sterile washcloth was saturated with 60ml of chlorhexidine gluconate (4%) cleansing solution and generously applied to the predefined surgical site followed by vigorous scrubbing for 3 min. (ii) after being patted with a sterile towel, the standardized 3-step disinfection was performed (iii) the applied iodine-alcohol disinfectant contained 70 ml of ethyl alcohol and 10 g of povidone-iodine per 100 ml
  Interventions: Drug: Chlorhexidine gluconate
- 0.9% Sodium Chloride ( N/S ) (Active Comparator): (i)a sterile washcloth was saturated with 60ml of sodium chloride (0.9%) and generously applied to the predefined surgical site followed by vigorous scrubbing for 3 min. (ii) after being patted with a sterile towel, the standardized 3-step disinfection was performed (iii) the applied iodine-alcohol disinfectant contained 70 ml of ethyl alcohol and 10 g of povidone-iodine per 100 ml
  Interventions: Drug: 0.9% Sodium Chloride

INTERVENTIONS:
Drug: Chlorhexidine gluconate — (i)a sterile washcloth was saturated with 60ml of chlorhexidine gluconate (4%) cleansing solution and generously applied to the predefined surgical site followed by vigorous scrubbing for 3 min. (ii) after being patted with a sterile towel, the standardized 3-step disinfection was performed (iii) the applied iodine-alcohol disinfectant contained 70 ml of ethyl alcohol and 10 g of povidone-iodine per 100 ml
  Other Names: Antigerm; Hibiscrub
  Arms: Chlorhexidine gluconate ( CHG )
Drug: 0.9% Sodium Chloride — (i)a sterile washcloth was saturated with 60ml of sodium chloride (0.9%) and generously applied to the predefined surgical site followed by vigorous scrubbing for 3 min. (ii) after being patted with a sterile towel, the standardized 3-step disinfection was performed (iii) the applied iodine-alcohol disinfectant contained 70 ml of ethyl alcohol and 10 g of povidone-iodine per 100 ml
  Other Names: normal saline
  Arms: 0.9% Sodium Chloride ( N/S )

SUMMARY:
To test whether pre - disinfection skin scrub with 4% chlorhexidine gluconate is more effective on the reduction of surgical site microbial colonization and subsequent infection than is normal saline.

DETAILED DESCRIPTION:
Surgical site infections (SSIs) following elective surgical procedures occur most commonly as a result of colonization by the patient's native skin flora . The most common pathogens causing SSIs are Staphylococcus aureus and coagulase-negative Staphylococci , components of normal skin flora . Therefore, preoperative disinfection of the surgical site with an antiseptic skin preparation is standard practice before any surgical intervention to decrease skin microbial counts before incision . It is considered an important step in limiting surgical wound contamination and preventing infection.

A variety of skin-preparation agents and methods are available for preventing surgical site infections and the techniques for preoperative cleansing of the skin vary among hospitals and surgeons. There is a pressing need to elucidate the effect of cutaneous disinfection with chlorhexidine gluconate ( CHG ) in prevention of surgical site infections.

Many studies demonstrated that comparisons with cutaneous disinfection with povidone-iodine, disinfection with CHG before insertion of an intravascular device and for post-infection site care can substantially reduce the incidence of device-related infection .

Hence, this study aimed to test whether an additional chlorhexidine gluconate scrub followed by a routine disinfection would lower the incidence of surgical site culture and subsequent infection after hepatic resection. This data will show the originality and clinical importance of a cutaneous pre-disinfection scrubbing solution for such risk patients with hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

* patient who received elective hepatectomy for liver tumors

Exclusion Criteria:

* patients who were younger than 18 years of age
* patients who had a history of radiation to the operative sites
* patients who received repeat hepatectomy
* patients who had a history of allergy to CHG, ethyl alcohol or povidone - iodine
* patients whose tumors were metastatic cancers
* patients who had a preoperative active remote infection

Ages: 18 Years to 92 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
the positive rate of the baseline culture , the preoperative culture , and the postoperative culture | within 30 days after the operation
  1. Before surgical preparation while the patient was on the table in the operating room , we obtained the first set of aerobic culture from the predefined incision site as the baseline culture.
  2. After skin scrubbing and disinfection , we obtained the second set of aerobic culture from the predefined incision site as the preoperative culture.
  3. After closure of the wound , we obtained the third set of aerobic culture from the surgical site as the postoperative culture.
  4. The result of culture was positive if bacteria were cultured from either stage of the surgical site sampling.
  5. We compared the efficacy for eradicating aerobic bacterial pathogens ( reduction of positive culture )from the abdomen between the chlorhexidine gluconate scrubbing group and normal saline scrubbing group .

SECONDARY OUTCOMES:
the post - operative surgical site infection | within 30 days after the operation
  Surgical site infection was using modified US Centers for Disease Control and Prevention definitions for nosocomial infection and documented by visiting patients everyday during the duration of hospitalization after surgery . After discharge , patients were checked weekly in the outpatient clinic to assess the surgical sites infection . All surgical site infections were classified as superficial , deep wound , or organ / space infection .
  We compared the incidence of post - operative surgical site infection between the chlorhexidine gluconate scrubbing group and normal saline scrubbing group .

CONTACTS AND LOCATIONS:
Overall Officials: YaoLi Chen, MD, Principal Investigator — Changhua Christian Hospital
Locations (1):
- Changhua Christian Hospital, Changhua, Changhua, Taiwan

REFERENCES:
- [Background] Noorani A, Rabey N, Walsh SR, Davies RJ. Systematic review and meta-analysis of preoperative antisepsis with chlorhexidine versus povidone-iodine in clean-contaminated surgery. Br J Surg. 2010 Nov;97(11):1614-20. doi: 10.1002/bjs.7214. PMID 20878942